CLINICAL TRIAL: NCT06524050
Title: Puppet Show and Storytelling Effect on Oral Medication Adherence and Negative Emotions Among Children With Cancer
Brief Title: Puppet Show and Storytelling Effect Among Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abeer Abd Elwahed Almowafy (Other)
Responsible Party: Sponsor-Investigator, Abeer Abd Elwahed Almowafy, Clinical Professor, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UB-RELOC H-06-BH-087)/ 1205.24
Record Dates: First submitted 2024-07-06; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Children With Cancer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puppet Show and Storytelling Effect among Children with Cancer (Experimental): puppet show and storytelling interventions
  Interventions: Behavioral: standard care
- standard care (No Intervention): standard care

INTERVENTIONS:
Behavioral: standard care — standard care
  Arms: Puppet Show and Storytelling Effect among Children with Cancer

SUMMARY:
Objective The objective of this study was to evaluate the effectiveness of puppet show and storytelling effect on oral medication adherence and negative emotions among children with cancer.

Methods A non-equivalent control group pre-test and post-test, between subjects design was conducted in the Maternity & Children Hospital Bisha, Al-Namas General Hospital, Kingdom of Saudi Arabia and Suez Canal University Hospital at Egypt. A total of 100 children (ages 3-12) admitted for treatments in this hospital were invited to participate in the study. Of the 100 paediatric patients; 50 received puppet show and storytelling interventions and 50 received usual care.

DETAILED DESCRIPTION:
Hospitalization is a stressful and threatening experience, which can be emotionally devastating to children with cancer. Pediatric nurses play interventions such as puppet show and storytelling have been used to promote oral medication adherence for children with cancer also to help them to overcome their negative emotions during hospitalization

.

ELIGIBILITY:
Inclusion Criteria:

* children with cancer who were diagnosed with the disease
* stay in the hospital for a minimum of three days in a row.
* The children were aged between three and twelve.

Exclusion Criteria:

* Children who were getting palliative care
* weren't enrolled in a comparable program
* those with recognized cognitive
* learning disabilities were not included in our sample

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Measurment tool: Questionnaire Evaluate the effectiveness of puppet shows and storytelling effect on oral medication adherence and negative emotions among children with cancer | 12 weeks
  Puppet Show and Storytelling Effect on Oral Medication Adherence and Negative Emotions among Children with Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Almowafy, Principal Investigator — Al-Azhar University
Locations (1):
- Abeer, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No